CLINICAL TRIAL: NCT01121367
Title: Study on Phenotypic Characterization of Combined Pulmonary Fibrosis and Emphysema
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: kewu Huang, MD, Beijing chaoyang hospital
Other Study IDs: KZ200910025007
Record Dates: First submitted 2010-05-06; First posted 2010-05-12 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-05

CONDITIONS: Pulmonary Fibrosis; Emphysema
Keywords: emphysema; pulmonary fibrosis;chemokine;sputum
MeSH Terms: conditions — Pulmonary Fibrosis; Emphysema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood, serum, sputum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Emphysema-alone
- CPFE group
- IPF-alone
- smokers
- nonsmokers

SUMMARY:
This study is to evaluate the expression of biological markers in induced sputum and peripheral blood T lymphocytes of patients with combined pulmonary fibrosis and emphysema (CPFE). The features of CPFE would be observed, including pulmonary function tests and fractional exhaled nitric oxide （FENO）.

DETAILED DESCRIPTION:
A new disease including concomitant upper-lobe emphysema and lower-lobe fibrosis in radiology has been defined as (combined pulmonary fibrosis and emphysema, CPFE). CPFE has distinct clinical characteristics with the emphysema and the pulmonary fibrosis, including gender, age, clinical manifestation, pulmonary function tests and prognosis.

Normally Th1/Th2 is balanced. However, patients with emphysema had a significantly higher expression of Th1. On the other hand, higher expression of Th2 is involved in the development of pulmonary fibrosis. The expressions of Th1 and Th2 were proved to play a central role in pathogenesis of emphysema and pulmonary fibrosis, while are still unknown in patients of combined pulmonary fibrosis and emphysema. The study would observe the Th1/Th2 expression, pulmonary function tests , fractional exhaled nitric oxide （FENO）and other features in CPFE patients.

ELIGIBILITY:
Inclusion Criteria:

1. IPF-alone group: 10 patients meeting the IPF diagnosis criteria without emphysema.
2. CPFE group: 15 patients with CT presentation of concomitant upper-lobe emphysema and lower-lobe fibrosis.
3. Emphysema-alone group: 15 patients with their CT diagnosis of emphysema without fibrosis.
4. Control: 20 healthy sex- and age-matched volunteers including nonsmokers and smokers. None of the healthy volunteers with a history of respiratory diseases.

Exclusion Criteria:

1. Age > 90 or < 50
2. Treated with corticosteroids or other immunomodulatory drugs
3. Some known causes of interstitial lung disease such as collagen vascular disease, drug-induced lung disease, occupational disease.
4. An exacerbation in 4 weeks
5. Subjects had a history of allergic diseases.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with emphysema，pulmonary fibrosis , combined pulmonary fibrosis and emphysema
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
the expression of CXCR3 in blood by flow cytometry and the chemokine IL-4,IFN-γ,CXCL9,CXCL10,CXCL11 and CCL17 in sputum and blood | six months

SECONDARY OUTCOMES:
pulmonary function tests | six months
fractional exhaled nitric oxide （FENO） | six months

CONTACTS AND LOCATIONS:
Overall Officials: kewu huang, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing chaoyang hospital-affiliate of captial medical university, Beijing, Beijing Municipality, China